CLINICAL TRIAL: NCT01913548
Title: Modulation of Iron Deposition in Sickle Cell Disease and Other Hemoglobinopathies SURVEY STUDY
Brief Title: Multi-Center Study of Iron Overload: Survey Study (MCSIO)
Acronym: MCSIO
Status: Completed | Type: Observational
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: University College London (UCL) Cancer Institute (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Medical University Innsbruck (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2010-019; 2R01DK057778-06A1 (NIH)
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Sickle Cell Disease; Thalassemia; Diamond-Blackfan Anemia
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia; Anemia, Diamond-Blackfan

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Sickle Cell Disease (SCD): Patients with sickle cell diseases, 16 years or older with 10-20 years of transfusion (defined as 0.2-0.6mg Fe/kg/day exposure with annual ferritin levels greater than 2500 in at least 60% of years of chronic transfusion); 0 to 9 years old at the initiation of chronic transfusions; no exchange transfusions in the previous 6 months; and iron overload documented by either liver biopsy, MRI or SQUID with estimated LIC (liver iron content) of greater than 7 mg/g dry wt in the previous 6 months or ferritin level greater than 1500mg/dl.
- Thalassemia Major (TM): Patients with β-thalassemia major and transfusion-dependent E-beta THAL. 16 years or older with 10-20 years of chronic transfusion (defined above), 0 to 9 years old at the initiation of chronic transfusions, iron overload documented by either liver biopsy, MRI or SQUID with estimated LIC of greater than 7 mg/g dry wt in the previous 6 months.
- Diamond Blackfan Anemia (DBA): Patients with DBA, 16 years or older with 10-20 years of transfusion, 0 to 9 years old at the initiation of chronic transfusions, iron overload documented by either liver biopsy, MRI or SQUID with estimated LIC of greater than 7 mg/g dry wt in the previous 6 months.

SUMMARY:
The purpose of this study is to demonstrate that a sufficient number of iron-overloaded thalassemia (THAL), Sickle Cell Disease (SCD)and Diamond Blackfan Anemia (DBA) populations with similar duration of chronic transfusion, and age at start of transfusions would be available for a confirmatory study. The study will examine the hypothesis that a chronic inflammatory state in SCD leads to hepcidin- and cytokine-mediated iron withholding within the RES (reticuloendothelial system), lower plasma NTBI (non-transferrin bound iron) levels, less distribution of iron to the heart in SCD.

DETAILED DESCRIPTION:
A detailed iron burden, transfusion and chelation history will be obtained from chart review or from participant recall.

Iron burden data will include: 1) documentation of liver iron, and 2) average annual ferritin values.

Transfusion data will include: (1) age at onset of regular transfusions, (2) years of chronic transfusion therapy, and (3) pre-transfusion Hb calculated as average of all assessments for each year.

ELIGIBILITY:
Inclusion Criteria:

* 10-20 years of transfusion (defined as 0.2-0.6mg Fe/kg/day exposure with annual ferritin levels greater than 2500 in at least 60% of years of chronic transfusion);
* 0 to 9 years old at the initiation of chronic transfusions; no exchange transfusions in the previous 6 months
* iron overload documented by either liver biopsy, MRI or SQUID with estimated LIC of greater than 7 mg/g dry wt in the previous 6 months or ferritin level greater than 1500mg/dl.

Exclusion Criteria:

* Patients with HbSC, HbS/β thalassemia
* Pacemaker (active or inactive) or other implanted magnetic devices, severe claustrophobia, or other contraindications to MRI; Unable to remove ferro-magnetic objects from the body in regions to be imaged (e.g., jewelry or piercing)
* Presence of any other condition which, in the opinion of the investigator, would make the patient unsuitable for enrollment;
* Any chronic inflammatory illness other than the SCD, THAL or DBA;
* Any acute illness within a 14 day period prior to blood sampling;
* Patients receiving intensive chelation in the 6 months prior to enrollment including deferoxamine 24 hours per day, 7 days per week or combination treatment with 2 chelators
* Pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: There is no gender predisposition for sickle cell disease, thalassemia major, or Diamond-Blackfan anemia. Sickle cell anemia most frequently affects people of African descent, thalassemia affects people of Mediterranian, northern African, Southeast Asia and Indian descent. Diamond-Blackfan anemia occurs across all racial and ethnic groups.
Sampling Method: Non-Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2010-03-31; Primary Completion 2013-08-31 (Actual); Study Completion 2013-10-31 (Actual)

PRIMARY OUTCOMES:
Identification of iron overloaded patients with Sickle Cell Disease and Thalassemia eligible for future study of iron deposition and biochemical mechanisms | March 2010 - July 2013
  Patients with similar duration of chronic transfusion and age at onset of chronic transfusion therapy will be identified from 10 participating centers. Detailed information on iron burden and transfusion, medical, and chelation histories will be obtained in order to establish a cohort of patients that could be available for a future powered study of extra-hepatic iron deposition and underlying biochemical mechanisms.

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Vichinsky, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland; John Porter, MD, Principal Investigator — University College London Cancer Institute
Locations (8):
- United States (6):
  - Children's Hospital & Research Center Oakland, Oakland, California
  - Georgia Regents University, Augusta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - Adult Comprehensive Sickle Cell Center, Duke University Medical Center, Durham, North Carolina
  - Thomas Jefferson SCD Program, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
- Universitätsklinikum Hamburg-Eppendorf, Hamburg-Eppendorf, Germany
- UCL Cancer Institute, London, United Kingdom